CLINICAL TRIAL: NCT01608308
Title: A Double Blind, Randomized, Placebo-controlled Study to Investigate the Effectiveness of IV Acetominophen Administered During Functional Endoscopic Sinus Surgery in Reducing the Use of Opiates to Treat Postoperative Pain
Brief Title: Intraoperative and Post-operative Analgesic Effect of IV Acetaminophen for Sinus Surgery
Acronym: IVAPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Davide Cattano, Associate Professor, Department of Anesthesia, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HSC-MS-12-0111
Record Dates: First submitted 2012-05-25; First posted 2012-05-31 (Estimated); Results first posted 2015-09-04 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Sinusitis
Keywords: Chronic Sinusitis; Pain Relief; Post-Operative Opioid Requirement; IV Acetaminophen; Functional Endoscopic Sinus Surgery; FESS
MeSH Terms: interventions — Acetaminophen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Acetaminophen (Experimental): The experimental group will receive a preoperative dose of 1000mg IV acetaminophen over 15 minutes. This will occur at least 15 minutes before the start of surgery. Another 1000mg dose of IV acetaminophen will be administered 4 hours after the first dose. A rescue analgesic containing oxycodone will also be provided (with APAP concentrations of 325 mg per Hospital and FDA recommendations).
  Interventions: Drug: IV Acetaminophen
- Control (Placebo Comparator): The control group (Placebo) will receive 100 mL of 0.9% normal saline in place of IV acetaminophen in the same manner as the experimental group; the investigator/physician in question will be blinded to the agent that is being administered. Patients will be discharged with instruction to continue APAP 500 mg PO every 6-8 hours. A rescue analgesic containing oxycodone will also be provided (with APAP concentrations of 325 mg per Hospital and FDA recommendations).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IV Acetaminophen — 1000mg IV acetaminophen over 15 minutes every 4 hours for up to 2 doses.
  Other Names: OFIRMEV (Cadence Pharamceutical, San Diego, USA)
  Arms: IV Acetaminophen
Drug: Placebo — 100 mL of 0.9% normal saline over 15 minutes in place of IV acetaminophen.
  Other Names: Normal Saline
  Arms: Control

SUMMARY:
The purpose of this study is to assess the use of IV acetaminophen (Ofirmev) as a and safe and efficacious agent in reducing post-operative pain; we hypothesize that its use will reduce post-operative pain when compared to a control group using the visual analogue score (VAS) analog pain scoring system.

DETAILED DESCRIPTION:
Unrelieved postoperative pain may result not only in suffering and discomfort, but may also lead to multiple physiological and psychological consequences which can contribute to adverse perioperative outcomes. Inadequate perioperative analgesia can potentially contribute to a higher incidence of myocardial ischemia. Additionally, the use of opioids has been associated with major side effects that can include impaired wound healing and delayed gastrointestinal (GI) motility that results in prolonged postoperative ileus.

Intravenous acetyl-para-aminophenol (APAP, also known as acetaminophen) is considered as the non-opioid analgesic of choice to treat postoperative mild and moderate pain, and has been demonstrated in several randomized trials to be both safe and effective at reducing acute post-operative pain in both children and adults. Furthermore, in the treatment of severe pain, it can reduce the need for opioid-analgesics while exhibiting a relatively limited side effect profile when compared to opioids and nonsteroidal anti-inflammatory drugs.

Chronic rhinosinusitis (CRS) describes a group of disorders characterized by inflammation of the nasal mucosa and/or paranasal sinuses for at least 12 consecutive weeks. In the United States, CRS affects approximately 30 million people, and represents 2% of the primary diagnoses in physician office visits, resulting in an estimated 200,000 sinus procedures annually. Patients suffering from CRS that is refractory to medical management complain of symptoms that include fatigue, headache, nasal drainage, facial pain and pressure, and decreased sense of smell. Functional endoscopic sinus surgery (FESS) represents a surgical approach to treating CRS that is unresponsive to medical management. Outcomes studies have identified FESS as efficacious at reducing the majority of symptoms related to CRS. Despite this, pain associated with CRS remains a significant co-morbidity that often is resistant to both medical and surgical management. Reducing the incidence and severity of acute post-operative pain is paramount to reducing the development of chronic pain that may exacerbate a patient's existing pain. The use of pre- and intra- operative IV acetaminophen thus serves as a unique pain management modality in this setting, as it has the potential for reducing post-operative complications and pain, with the additional benefit of minimal intraoperative bleeding, an undesirable complication often associated with FESS and with the use of non-steroidal anti-inflammatory drugs (NSAIDs).

The use of IV acetaminophen in ear, nose, and throat (ENT) surgery is not a novel endeavor. Indeed, studies have demonstrated the efficacy and safety of IV acetaminophen for use in tonsillectomy and FESS. We wish to provide a more comprehensive analysis of pain management in the setting of FESS in the following ways :

1. by administering IV acetaminophen perioperatively (before start of surgery, and after surgery completion;
2. by employing a pain score of 4 (whereas other studies use 3) as a cutoff for breakthrough pain; and,
3. by addressing novel outcomes including patient sedation and patient satisfaction, in addition to opioid analgesic use.

In our institution, we have completed a preliminary pilot study exploring the use of intravenous anesthesia which included acetaminophen during bilateral endoscopic sinus surgery. Secondary outcomes measured during the study included:

1. Pain
2. Rescue analgesic use
3. Nausea/Vomiting
4. Time spent in recovery
5. Successful discharge from the PACU and the Hospital

Our pilot data has reaffirmed that the procedure is overall benign, with few associated risks and adverse events. Of note, none of the patients in our preliminary study required admission to the hospital after surgery for further observation as a result of uncontrolled pain or nausea. Based on this experience, we would like to explore the efficacy of intravenous acetaminophen (Ofirmev), a non opioid/non steroidal analgesic, in endoscopic sinus surgery.

ELIGIBILITY:
Inclusion criteria:

1. Patients undergoing surgical management for CRS (with or without polyps)
2. Operating time must be at least 2 hours in duration.
3. Number of sinuses involved must be 3 or greater

Exclusion criteria:

1. History of hypersensitivity to acetaminophen
2. End stage renal disease
3. End stage liver disease
4. History of chronic pain, or use of opioid medication in the previous two weeks
5. Severe depression or anxiety
6. Use of gabapentin or any other pain modulator
7. History of acute sinusitis or mucocele
8. History of seizures
9. Known or suspected history of alcohol or drug abuse
10. Known or suspected history of morphine intolerance

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Cattano, MD, PhD, Principal Investigator — The University of Texas Health Sciences Center at Houston
Locations (1):
- The University of Texas Health Sciences Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Tyler MA, Lam K, Ashoori F, Cai C, Kain JJ, Fakhri S, Citardi MJ, Cattano D, Luong A. Analgesic Effects of Intravenous Acetaminophen vs Placebo for Endoscopic Sinus Surgery and Postoperative Pain: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2017 Aug 1;143(8):788-794. doi: 10.1001/jamaoto.2017.0238. PMID 28542675

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment is completed.
Groups:
- IV Acetaminophen: The experimental group will receive a preoperative dose of 1000mg IV acetaminophen over 15 minutes. This will occur at least 15 minutes before the start of surgery. Another 1000mg dose of IV acetaminophen will be administered 4 hours after the first dose. A rescue analgesic containing oxycodone will also be provided (with acetyl-para-aminophenol (APAP, also known as acetaminophen) concentrations of 325 mg per Hospital and FDA recommendations).
  IV Acetaminophen: 1000mg IV acetaminophen over 15 minutes every 4 hours for up to 2 doses.
- Control: The control group (Placebo) will receive 100 mL of 0.9% normal saline in place of IV acetaminophen in the same manner as the experimental group; the investigator/physician in question will be blinded to the agent that is being administered. Patients will be discharged with instruction to continue APAP 500 mg PO every 6-8 hours. A rescue analgesic containing oxycodone will also be provided (with acetyl-para-aminophenol (APAP, also known as acetaminophen) concentrations of 325 mg per Hospital and FDA recommendations).
  Placebo: 100 mL of 0.9% normal saline over 15 minutes in place of IV acetaminophen.
Period: Overall Study
Arm/Group | IV Acetaminophen | Control
Started | 31 | 31
Completed | 31 | 29
Not Completed | 0 | 2
Not completed — pretreatment medical and billing reasons | 0 | 2

BASELINE CHARACTERISTICS:
Population: In total 62 subjects were enrolled. Two subjects were dropped due to pretrreatment medical and billing issues;therefore, in total 60 subjects were dosed.
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Acetaminophen | Control | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (14.6) | 54.2 (14.4) | 53.95 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 17 | 26
  Male | 22 | 14 | 36
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Pain Level Assessed Using a Visual Analogue Scale (VAS) Scale
Description: VAS is a validated, self-reported data sheet assessing average pain intensity. Possible scores range from 0 (no pain) to 10 (highest level of pain).
Time Frame: 15 minutes and 120 minutes Post-Operatively
Population: At the 15 minute time point, data was obtained for 24 participants in the acetaminophen group and 26 participants in the control group. For the 120 minute time point, data was obtained for 7 participants in the acetaminophen group and 11 participants in the control group.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | IV Acetaminophen | Control
Number analyzed (Participants) | 24 | 26
units on a scale
  15 minutes (n=24, 26) | 0 [0 to 3] | 0 [0 to 4]
  120 minutes (n=7, 11) | 0 [0 to 2] | 2 [0 to 4]

2. Secondary Outcome: Total Doses of Postoperative Opiate (Morphine) Use
Description: The total amount of morphine utilized in Postoperative Acute Care Unit (PACU) will be recorded. One dose is a 1mg bolus of morphine.
Time Frame: During Postoperative Acute Care Unit (PACU) stay (up to 4 hours after surgery)
Measure: Median (Inter-Quartile Range); unit: doses
Arm/Group | IV Acetaminophen | Control
Number analyzed (Participants) | 31 | 29
doses | 1.5 [1 to 2.5] | 2.5 [2 to 4]

3. Secondary Outcome: Number of Participants Who Received Intraoperative Supplemental Fentanyl
Description: Number of participants who received intraoperative supplemental fentanyl. The decision to administer fentanyl is based on hemodynamic changes, such as increasing blood pressure and heart rate.
Time Frame: During Postoperative Acute Care Unit (PACU) stay (up to 4 hours after surgery)
Measure: Number; unit: participants
Arm/Group | IV Acetaminophen | Control
Number analyzed (Participants) | 31 | 29
participants | 9 | 4

4. Secondary Outcome: Number of Participants Who Experienced Postoperative Morbidity (Nausea)
Description: Post-operative nausea will be monitored and measured through direct observation and nursing clinical record
Time Frame: During Postoperative Acute Care Unit (PACU) stay (up to 4 hours after surgery)
Measure: Number; unit: participants
Arm/Group | IV Acetaminophen | Control
Number analyzed (Participants) | 31 | 29
participants | 13 | 10

5. Secondary Outcome: Postoperative Vital Sign (Systolic Blood Pressure)
Description: Postoperative vital signs (systolic and diastolic blood pressure, pulse, temperature, and respiratory rate) were measured at different time points up to 4 hours after surgery.
Time Frame: During Postoperative Acute Care Unit (PACU) stay (up to 4 hours after surgery)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | IV Acetaminophen | Control
Number analyzed (Participants) | 28 | 27
mmHg | 133 (17.2) | 144 (15)

6. Secondary Outcome: Postoperative Vital Sign (Diastolic Blood Pressure)
Description: as for outcome 5
Time Frame: During Postoperative Acute Care Unit (PACU) stay (up to 4 hours after surgery)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | IV Acetaminophen | Control
Number analyzed (Participants) | 28 | 27
mmHg | 75 (13.5) | 78.3 (10.5)

7. Secondary Outcome: Postoperative Vital Sign (Pulse)
Description: as for outcome 5
Time Frame: During Postoperative Acute Care Unit (PACU) stay (up to 4 hours after surgery)
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | IV Acetaminophen | Control
Number analyzed (Participants) | 29 | 27
beats per minute | 76.3 (12.4) | 80 (13.2)

8. Secondary Outcome: Postoperative Vital Sign (Temperature)
Description: as for outcome 5
Time Frame: During Postoperative Acute Care Unit (PACU) stay (up to 4 hours after surgery)
Measure: Mean (Standard Deviation); unit: Fahrenheit
Arm/Group | IV Acetaminophen | Control
Number analyzed (Participants) | 29 | 26
Fahrenheit | 97.1 (0.8) | 97.4 (0.8)

9. Secondary Outcome: Postoperative Vital Sign (Respiratory Rate)
Description: as for outcome 5
Time Frame: During Postoperative Acute Care Unit (PACU) stay (up to 4 hours after surgery)
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | IV Acetaminophen | Control
Number analyzed (Participants) | 31 | 29
breaths per minute | 17.4 (1.2) | 17.2 (1.3)

ADVERSE EVENTS:
Arm/Group | IV Acetaminophen | Control
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 13/31 | 10/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV Acetaminophen (N=31) | Control (N=29)
Nausea (Surgical and medical procedures) | 13 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No